CLINICAL TRIAL: NCT01176292
Title: A Prospective Comparison of Rotating Platform Cruciate Substituting Total Knee Arthroplasty With Rotating Platform High-Flex Cruciate Substituting Total Knee Arthroplasty
Brief Title: Comparison of High Flex and Standard Rotating Platform Total Knee Arthroplasty (TKA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anderson Orthopaedic Research Institute (Other)
Collaborators: DePuy Orthopaedics (Industry)
Responsible Party: Principal Investigator, William G. Hamilton, MD, Principal Investigator, Anderson Orthopaedic Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AORI2010-0104
Record Dates: First submitted 2010-07-26; First posted 2010-08-06 (Estimated); Results first posted 2015-08-31 (Estimated); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Knee Osteoarthritis
Keywords: total knee replacement; high flexion; range of motion; rotating platform; TKA
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rotating Platform High-Flex Cruciate Substituting TKA (Other)
  Interventions: Device: Rotating Platform High-Flex Cruciate Substituting TKA
- Rotating Platform Cruciate Substituting TKA (Other)
  Interventions: Device: Rotating Platform Cruciate Substituting TKA

INTERVENTIONS:
Device: Rotating Platform High-Flex Cruciate Substituting TKA
  Arms: Rotating Platform High-Flex Cruciate Substituting TKA
Device: Rotating Platform Cruciate Substituting TKA
  Arms: Rotating Platform Cruciate Substituting TKA

SUMMARY:
The goal of this study is to determine if the rotating platform high flex design provides improved flexion compared to the standard rotating platform TKA.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 75 years old
* Primary diagnosis of osteoarthritis of the knee
* Patients who, in the investigator's opinion, are appropriate candidates for a cemented, rotating platform TKA.
* Patients who, in the investigator's opinion, are capable of participation in a clinical trial and reliable enough to return for follow-up appointments.

Exclusion Criteria:

* Pregnant or lactating female subjects
* Patients with post-traumatic or inflammatory arthritis
* Patients with a fixed flexion contracture of greater than 20 degrees
* Patients with advanced hip, spine, or ankle disease
* Patients with a BMI greater than 40, where knee flexion may be limited by soft tissues

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2007-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William G Hamilton, MD, Principal Investigator — Anderson Orthopaedic Research Institute

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject enrollment began August 2007 and ended April 2009, with a total of 142 patients enrolled at an orthopaedic clinic.
Period: Overall Study
Arm/Group | Rotating Platform High-Flex Cruciate Substituting TKA | Rotating Platform Cruciate Substituting TKA
Started | 71 | 71
Completed | 66 | 62
Not Completed | 5 | 9
Not completed — Lost to Follow-up | 2 | 4
Not completed — Adverse Event | 1 | 1
Not completed — Physician Decision | 0 | 2
Not completed — Has not scheduled one-year visit yet | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rotating Platform High-Flex Cruciate Substituting TKA | Rotating Platform Cruciate Substituting TKA | Total
Number analyzed (Participants) | 71 | 71 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (7) | 62 (7) | 64 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 44 | 81
  Male | 34 | 27 | 61

OUTCOME MEASURES:

1. Primary Outcome: Clinical Flexion
Description: Maximum, passive flexion and extension of the operated knee joint in the supine position will be measured and recorded using a long goniometer.
Time Frame: Preoperative, 4-6 weeks
Population: All subjects with available data at the preoperative and 4-6 week intervals.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Rotating Platform High-Flex Cruciate Substituting TKA | Rotating Platform Cruciate Substituting TKA
Number analyzed (Participants) | 70 | 68
degrees
  Clinical flexion - preoperative | 119.1 (13.2) | 120.3 (11.2)
  Clinical flexion - 4 week | 112.0 (12.7) | 111.3 (15.3)

2. Secondary Outcome: Radiographic Flexion
Description: Lateral radiographs of the knee will be taken with the patient supine with maximal passive knee flexion. Flexion will then be measured directly from these radiographs.
Time Frame: preoperative, 4-6 weeks
Population: All subjects with available data at the preoperative and 4-6 week intervals.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Rotating Platform High-Flex Cruciate Substituting TKA | Rotating Platform Cruciate Substituting TKA
Number analyzed (Participants) | 70 | 68
degrees
  preoperative | 116.8 (14.1) | 116.6 (15.5)
  4-6 weeks | 104.7 (16.3) | 102.1 (16.4)

3. Secondary Outcome: Radiographic Flexion
Description: as for outcome 2
Time Frame: 1 year
Population: All subjects with available data at the 1-year interval.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Rotating Platform High-Flex Cruciate Substituting TKA | Rotating Platform Cruciate Substituting TKA
Number analyzed (Participants) | 66 | 62
degrees | 117.6 (11.1) | 117.9 (11.6)

4. Secondary Outcome: Knee Society Score (KSS)
Description: A standard clinical evaluation system for reporting results for patients undergoing total knee replacement. The minimum score is 0 and the highest score is 100. A higher score represents a better outcome.
Time Frame: 1 year
Population: All subjects with available KSS data at the 1-year interval.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Rotating Platform High-Flex Cruciate Substituting TKA | Rotating Platform Cruciate Substituting TKA
Number analyzed (Participants) | 66 | 62
score
  Clinical KSS | 95.0 (8.4) | 94.9 (8.3)
  Functional KSS | 87.7 (19.9) | 90.9 (16.0)

5. Secondary Outcome: Oxford Knee Score
Description: A patient reported questionnaire for assessing the outcome of knee surgery. The minimum score is 0 and the maximum score is 48. A higher score represents a better outcome.
Time Frame: 1 year
Population: All subjects with available Oxford Knee Score data at the 1-year interval.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Rotating Platform High-Flex Cruciate Substituting TKA | Rotating Platform Cruciate Substituting TKA
Number analyzed (Participants) | 59 | 57
score | 41.0 (6.5) | 41.8 (7.4)

6. Primary Outcome: Clinical Flexion
Description: as for outcome 1
Time Frame: 4-6 months
Population: All subjects with available data at the 4-6 month interval.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Rotating Platform High-Flex Cruciate Substituting TKA | Rotating Platform Cruciate Substituting TKA
Number analyzed (Participants) | 70 | 65
degrees | 122.5 (8.6) | 121.3 (9.6)

7. Primary Outcome: Clinical Flexion
Description: as for outcome 1
Time Frame: 1 year
Population: All subjects with available data at the 1-year interval.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Rotating Platform High-Flex Cruciate Substituting TKA | Rotating Platform Cruciate Substituting TKA
Number analyzed (Participants) | 66 | 62
degrees | 124.2 (8.7) | 124.0 (10.3)

ADVERSE EVENTS:
Time Frame: 1 year follow-up
Description: Collected according to standard protocol.
Arm/Group | Rotating Platform High-Flex Cruciate Substituting TKA | Rotating Platform Cruciate Substituting TKA
Serious Adverse Events (participants affected / at risk) | 7/71 | 4/71
Other Adverse Events (participants affected / at risk) | 9/71 | 3/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotating Platform High-Flex Cruciate Substituting TKA (N=71) | Rotating Platform Cruciate Substituting TKA (N=71)
infection (Infections and infestations) | 1 (1) | 1 (1) — Infection/polyethylene exchange
stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) — manipulation for stiffness
patellar fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Repair of patellar fracture due to a fall.
quadriceps tendon rupture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Extensor mechanism reconstruction from a quadriceps tendon rupture.
symptomatic patellar crepitus (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) — Arthroscopic nodule debridement for patellar crepitus
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotating Platform High-Flex Cruciate Substituting TKA (N=71) | Rotating Platform Cruciate Substituting TKA (N=71)
postoperative pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
patellar crepitus (Musculoskeletal and connective tissue disorders) | 9 (9) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any paper drafted by authors regarding project results should be sent to sponsor at least 30 days before being submitted for publication. An abstract should be sent to the sponsor at least 10 days before being submitted. The sponsor will inform the authors of any changes deemed necessary to preserve the confidentiality of proprietary information or to insure scientific accuracy.